CLINICAL TRIAL: NCT03613675
Title: Acceptability of Video Games to Promote Asthma Education and Self-management in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Concordia University, Montreal (Other)
Responsible Party: Principal Investigator, Sze Man Tse, Assistant professor, pediatric respirologist, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2019-2075
Record Dates: First submitted 2018-07-27; First posted 2018-08-03 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Asthma
Keywords: video games
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Participants will be asked to play 4 video games on asthma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video games (Experimental): All participants will be asked to play 4 video games.
  Interventions: Device: Video games

INTERVENTIONS:
Device: Video games — The 4 videos games consists of:
  * Asthmonaut, a desktop game in which the child navigates through different scenarios and interacts with nine characters to learn about asthma symptoms and management (30 minutes)
  * Lung Launcher, a mobile game in which the character encounters different asthma triggers (customizable to the child) and the child has to find the correct preventive method to address each trigger (4 minutes)
  * Asthma Heroes, a desktop game where the player interacts with several characters to learn about their symptoms, treatment and context, and collects objects to help them manage their asthma (30 minutes)
  * Bloïd, a mobile game where the player uses a pressure sensor as an input device to guide a spacecraft and destroy meteorites in its path (4 minutes).

SUMMARY:
Asthma is a chronic lung disease affecting over 800,000 Canadian children. Knowing how to avoid asthma triggers, to take care of one's health, and to know when and why to do one's treatment can help prevent asthma crises, and have a better quality of life.

Games in health can make the management of asthma easier by helping the child better understand his condition, his triggers, and manage his asthma by himself. Games also offer a personalized experience, where players can receive feedback about their learning. However, few studies explored the use of games in childhood asthma.

This study will test 4 games for children with asthma. Through different characters and scenarios, the goals of the games are to help the child with asthma to better recognize and manage his asthma triggers and symptoms. The objectives of this study are:

* Evaluate the acceptability of these games in children with asthma
* Gather feedback on the games to guide future development

ELIGIBILITY:
Inclusion Criteria: Along with a parent, children

* aged 8-12 years inclusively
* with physician-diagnosed asthma
* who are on a daily controller medication
* who understand French or English.

Exclusion Criteria: children with

* chronic respiratory conditions other than asthma
* cardiovascular diseases
* neuromuscular disorders
* developmental delay.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Gaming experience, relevance for end-user, and areas of improvement of the games | Immediately after playing the games (same day)
  This is a qualitative outcome which includes the quality of the interface as assessed by the player, the gaming experience, its relevance for the end-user, and areas of improvement. This will be assessed through a questionnaire and a focus group.

SECONDARY OUTCOMES:
Asthma knowledge | Immediately after playing the games (same day)
  This includes retention of key messages and whether the games respond to the families' knowledge gaps. Knowledge transfer will be assessed through a questionnaire administered to the child before and after the gaming experience. This questionnaire contains 16 true or false questions and 5 questions with short answers on asthma. The maximal score on this questionnaire is 25 (range 0-25).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No